CLINICAL TRIAL: NCT06745401
Title: Remote Monitoring of Cancer Patients With Outpatient Treatment
Status: Completed | Type: Observational
Sponsor: Persei Vivarium (Other)
Collaborators: Effice Servicios Para la Investigacion S.L. (Industry)
Responsible Party: Sponsor
Other Study IDs: PersV.Onco.DTx01
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Cancer Patients With Outpatient Treatment
Keywords: Remote patient monitoring; Cancer patients; outpatient treatment; Caaring; real-world data; DTx; patient-reported data; Digital Health; PROMs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This project focuses on studying the use of digital platforms for monitoring, between medical visits, parameters such as toxicities and therapeutic adherence.

The goal of this observational study is to know the degree of usability of the Caaring® digital platform in cancer patients undergoing outpatient oral treatment. This will allow in the future to design comparative studies that demonstrate the advantages of using this application in the management of these patients.

Participants will fill out various questionnaires in the Caaring app related to their symptoms, adherence to treatment, quality of life and physical activity, among others.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients with adjuvant or metastatic oncological treatment
* Cancer patients with oral oncological treatment
* Patients who are able to complete the study questionnaires
* Patients who are able to handle the application on a smart mobile phone.
* Informed consent is obtained from the patient.

Exclusion Criteria:

* Patients who will not be able to commit to carrying out the follow-ups or do not have adequate technological skills.
* Patients with inability to give adequately the informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cancer Patients from the Hospital HM Sanchinarro diagnosed who meet the selection criteria and sign the informed consent will be included.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2024-11-21 (Actual); Primary Completion 2025-03-03 (Actual); Study Completion 2025-03-03 (Actual)

PRIMARY OUTCOMES:
Usability of Caaring® for the management of oncology patients in outpatient oral treatment | Day 0 up to 3 months
  Percentage of patients with at least 80% of the data completed in the application, Percentage of patients with 100% of the data completed in the application and Percentage of completion per patient

SECONDARY OUTCOMES:
Degree of completion of data relating to treatment adherence | Weekly up to 3 months
  The Degree of completion of therapeutic adherence by patients in Caaring application between visits is defined as the ratio between the questionnaires requested and completed.
Degree of completion of data related to the toxicity of their treatment | Weekly up to 3 months
  The Degree of completion of toxicity of their treatments by patients in Caaring application between visits: Percentage of patient participation defined as data completed among requested data; Percentage of patients with at least 80% of the data completed; Percentage of patients with 100% of the data completed and Percentage of patients with at least 80% of the data completed by questionnaire
Quality of the care process through impact on the patient's quality of life: WHOQOL | Day 0 and week 12
  Changes in patient's quality of life scale WHOQOL (World Health Organization Quality of Life) scores at the end of the study compared to baseline. Values (0-100), a higher score reflects a higher health-related quality of life.
Quality of the care process through impact on the patient's quality of life: IPAQ | Day 0 and week 12
  Changes in International Physical Activity Questionaire (IPAQ) scores at the end of the study compared to baseline. Values (46-100), a higher score reflects a higher Physical Activity
Patient workload | Week 12
  Evaluate the Patient workload through the percentage of patients who complete the study correctly by completing all questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital HM Sanchinarro, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No